CLINICAL TRIAL: NCT04810689
Title: A Randomized, Double-Blind, Placebo-Control Pilot Trial of Xuanfei Baidu Granules (XFBD), a Traditional Chinese Medicine (TCM), in Persons With COVID-19
Brief Title: Pilot Trial of XFBD, a TCM, in Persons With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futile Enrollment
Sponsor: Darcy Spicer (Other)
Responsible Party: Sponsor-Investigator, Darcy Spicer, Associate Professor, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HS-20-00632
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Covid19
Keywords: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to 1 of 2 arms: XFBD granules or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XFBD Arm (Experimental): XFBD (administered as 1 packet of granules dissolved in warm water) orally twice daily for 14 day, 1 hour after food in the morning and at night with at least 8 hours in between doses
  Interventions: Drug: Xuanfei Baidu Granules
- Placebo Arm (Placebo Comparator): Placebo (administered as 1 packet of granules dissolved in warm water) orally twice daily for 14 day, 1 hour after food in the morning and at night with at least 8 hours in between doses
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Xuanfei Baidu Granules — Xuanfei Baidu granules is a prescription of 13 herbal medicinals made into dissolvable granules for oral intake
  Other Names: XFBD
  Arms: XFBD Arm
Other: Placebo — Placebo for Xuanfei Baidu granule made into dissolvable granules for oral intake
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to document the safety of taking traditional Chinese medicine (TCM) in patients with COVID-19 and to gain information to determine whether a study with TCM can be conducted. The study will test a traditional Chinese medicine that has been made into a granule formulation called Xuanfei Baidu Granules.

DETAILED DESCRIPTION:
Xuanfei Baidu granules (XFBD) is a 13 medicinal traditional Chinese medicine (TCM) prescription developed by Dr. Zhang Boli, a member of Chinese Academy of Engineering, and his team, and used in Wuhan, China, during the initial outbreak of SARS-CoV2. Based on TCM theory, the 13 medicinals used mainly consist of heat-clearing and toxin-removing medicinals to reduce fever and clear viruses; cough-suppressing and phlegm-transforming medicinals to thin and clear the phlegm; and lung-diffusing and pant-calming to soothe the tracheal smooth muscle and relieve shortness of breath. Another unique quality is one of the medicinals helps to dissipate stasis and dissolves blood clots, providing a mild anticoagulant effect.

Before the widespread usage of TCM, nationwide China saw a progression of disease of about 10% of their mild and moderate cases while during the period with the TCM utilization, the percentage dropped to 2-5% depending on the hospital. Overall, they saw an improvement of clinical symptoms. Due to the challenges of the rapidly evolving outbreak, these are clinical observations and not evidence from a controlled study.

The purpose of this initial pilot study is to document the safety of taking a TCM in patients with COVID-19 and to gain information to determine whether a study with TCM can be conducted in the US. The study will test a TCM which has been made into a granule formulation called XFBD.

This is a randomized double-blind placebo-control pilot trial to document safety and efficacy endpoint assessments and to determine the feasibility of community recruitment and enrollment of symptomatic adult outpatients with COVID-19. The 12-week pilot will have 14 days where they receive XFBD or a placebo, orally twice a day and a 10 week follow up. The study will have a total of 60 participants with approximately 30 participants in each treatment arm. The participants will be randomized 1:1 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participant provides informed consent prior to initiation of any study procedures.
* Individual 18 to 75 years of age.
* Documentation of confirmed active SARS-CoV-2 infection, as determined by an FDA authorized molecular test conducted at any US clinic or laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent from any respiratory specimen collected <96 hours prior to study entry.
* Mild or Moderate COVID-19 experiencing at least one SARS-CoV-2 infection symptom including:

  * Mild Covid-19: Symptoms of mild illness with COVID-19 that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea
  * Moderate Covid-19:

    * Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion
    * Presence of clinical signs consistent with moderate illness with COVID-19, such as respiratory rate ≥ 20 breaths per minute, saturation of oxygen (SpO2) > 93% on room air at sea level, heart rate ≥ 90 beats per minute from a health care encounter within 48 hours.
* Agrees to not participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 during the study period up until reaching hospitalization or 28 days, whichever is earliest.
* Agrees to not utilize TCM outside of this study.
* Willing to be randomized to XFBD and placebo control arm for 14 days, and followed up to 12 weeks.
* Willing to comply with the study related questionnaires, procedures and measurements.
* Will to not become pregnant during the 14 days of test substance ingestion using appropriate accepted methods of contraception. Acceptable methods of contraception include: postmenopausal 1 year of amenorrhea and over 50 years of age; prior tubal ligation or hysterectomy; or barrier contraception using condom or diaphragm plus spermicide.
* Able to provide the identity of their health care provider or health system clinical care entry information.
* Able to utilize telephone and telehealth platform to comply with the study related questionnaires, procedures and measurements. Established during the recruitment process.
* Able to speak and communicate in English, Spanish, Mandarin Chinese or Cantonese.

Exclusion Criteria:

* Need for hospitalization.
* Severe or Critical COVID-19:

  * Severe COVID-19

    * Symptoms suggestive of severe systemic illness with COVID-19, which could include any symptom of moderate illness or shortness of breath at rest, or respiratory distress
    * Clinical signs indicative of severe systemic illness with COVID-19, respiratory rate ≥ 30 breaths per minute, heart rate ≥ 125 beats per minute, SpO2 ≤ 93% on room air at sea level or respiratory PaO2/FiO2 < 300
  * Critical COVID-19 -- Evidence of critical illness, defined by at least one of the following:

    * Respiratory failure defined based on resource utilization requiring at least one of the following: Endotracheal intubation and mechanical ventilation, oxygen delivered by high flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation)
    * Shock (defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg or requiring vasopressors)
    * Multi-organ dysfunction/failure
* Positive SARS-CoV-2 molecular test in the absence of Covid-19 symptoms. However if patients develop symptoms within 14 days of the positive test and fulfill all other enrollment criteria, they are eligible for participation.
* Receiving the following classes of agents found in 5.4.1. Prohibited Medications
* Use of drugs for anti-SARS-CoV-2 treatment including remdesivir, baricitinib, lopinavir/ritonavir fixed dose combination, ribavirin, chloroquine, hydroxychloroquine, and azithromycin, dexamethasone, bamlanivimab, casirivimab plus imdevimab convalescent plasma, or participation in a clinical trial involving any of these drugs whether for treatment or prophylaxis.
* Participating in a study where co-enrollment is not allowed.
* Receipt of a SARS-CoV-2 vaccination prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of XFBD
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Has known prior kidney disease.
* Has known cirrhosis, acute liver disease or uncontrolled chronic liver disease.
* Has known severe coronary artery disease.
* Has known narrow angle glaucoma.
* Has greater than two or a single uncontrolled underlying comorbid condition including cardiovascular disease (coronary artery disease, heart failure, valvular heart disease), hypertension, diabetes, chronic lung disease, chronic kidney disease, chronic liver disease, immunocompromised (HIV or daily users of more than 5 mg/day of prednisone), prior organ transplant.
* Fulfills the FDA EUA criteria of at high risk for progressing to severe COVID-19. This includes high-risk individuals specified in the EUA who meet at least one of the following criteria: Body mass index (BMI) ≥35; Chronic kidney disease; Diabetes mellitus; Immunocompromising condition/immunosuppressive disease; Currently receiving immunosuppressive treatment; Aged ≥65 years; or Aged ≥55 years and have: Cardiovascular disease, or Hypertension, or Chronic obstructive pulmonary disease/other chronic respiratory disease. If the patient is not able to receive the EUA agent casirivimab and imdevimab (Regeneron) or bamlanivimab (Eli Lilly) because of unavailability this exclusion may be waived.
* Women who are currently pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy V Spicer, MD, Principal Investigator — Keck Medicine of USC
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using a COVID-19 registry at the time of testing in Los Angeles County between March 2021 through June 2022. A total 10 individuals consented and 5 were randomized and received study medication. The first participant was enrolled March 2021 and the last participant was enrolled February of 2022. The study was terminated for futility.
Pre-assignment Details: Of the 10 subjects who consented 5 were randomized and 5 withdrew before randomization.
Period: Overall Study
Arm/Group | XFBD Arm | Placebo Arm
Started | 3 | 2
Completed | 3 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XFBD Arm | Placebo Arm | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Agreement to Participate
Description: To document the proportion of patients who agree to participate as measured by enrollment and randomization.
Time Frame: 15.5 months
Population: Enrollment insufficient and hence trial terminated.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled: Patients who expressed interest in participating and signed the informed consent
Arm/Group | Enrolled
Number analyzed (Participants) | 10
Participants
  Randomized into XFBD Arm | 3
  Randomized into Placebo Arm | 2
  Did not start study | 5

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | XFBD Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XFBD Arm (N=3) | Placebo Arm (N=2)
insomnia (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study failed to enter a sufficient number of subjects for any meaningful analysis and was terminated for futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04810689/Prot_SAP_ICF_001.pdf